CLINICAL TRIAL: NCT03788538
Title: Effects of Dexmedetomidine on Modulation of Perioperative Blood Glucose and Related Hormones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhuan Zhang, Clinical Professor, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20181224
Record Dates: First submitted 2018-12-25; First posted 2018-12-27 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Dexmedetomidine; Blood Glucose
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group 1 with no dexmedetomidine (No Intervention)
- group 2 with dexmedetomidine 0.25μg/kg/h (Experimental)
  Interventions: Drug: dexmedetomidine
- group 2 with dexmedetomidine 0.5μg/kg/h (Experimental)
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — 10 minutes before anesthesia induction, all patients were administrated with dexmedetomidine 1 μg/kg/min.At the beginning of induction, dexmedetomidine was changed to corresponding maintenance dose in each group.
  Arms: group 2 with dexmedetomidine 0.25μg/kg/h; group 2 with dexmedetomidine 0.5μg/kg/h

SUMMARY:
The investigators aimed to explore effects of dexmedetomidine on modulation of perioperative blood glucose and relevant hormone during the general anesthesia with surgery time ≥ 4 hours, and the effects on postoperative complications. 75 participants (American Society of Anesthesiologists grades I or II, of both sexes,aged 40-80 yr,with BMI of 18.5-27 kg/m2) scheduled for elective surgery under general anesthesia with surgery time ≥ 4 hours were enrolled in this study. The participants were divided into four groups: group C (control saline group, no dexmedetomidine use), group D1 (dexmedetomidine loading dose 1 mcg/kg, maintenance dose 0.25 mcg/kg/h), group D2 (dexmedetomidine loading dose 1 mcg/kg, maintenance dose 0.5 mcg/kg/h).10 minutes before anesthesia induction, all participants were administrated with dexmedetomidine 1 μg/kg/min.At the beginning of induction, dexmedetomidine was changed to corresponding maintenance dose in each group. Blood samples were taken at the beginning of dexmedetomidine (T0), the beginning of skin incision (T1), 1 h after skin incision (T2), the end of the surgery (T3) and 1 h after patient transfer to PACU (T4) for the value of blood glucose,lactate and relevant hormones. Also, investigators also record the total amount of propofol and sufentanil at the end of surgery,and the complications within 24 h after the surgery.

ELIGIBILITY:
Inclusion Criteria:

- patients undergoing operations over 4 h under general anesthesia,ASA physical status I or II, irrespective of showing gender bias, aged between 50-75 years old, and having a body mass index (BMI) between 18.5-28 kg/m2.

Exclusion Criteria:

* the patients with bradycardia, hypoglycemia, heart disease, adrenal tumor,diabetes or showed ≥7.0 mmol/L, or HbA1c level ≥6.5%.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Effects of dexmedetomidine on perioperative blood glucose (mmol/L) | before dexmedetomidine infusion, 1 hour after incision, at the end of surgery, 1 hour after patient transfer to postanesthesia care unit..
  The changes of blood glucose during the surgery period
Effects of dexmedetomidine on perioperative insulin (μIU/ml) | before dexmedetomidine infusion, 1 hour after incision, at the end of surgery, 1 hour after patient transfer to postanesthesia care unit.
  The changes of insulin during the surgery period
Effects of dexmedetomidine on perioperative glucagon and catecholamine (pg/ml) | before dexmedetomidine infusion, 1 hour after incision, at the end of surgery, 1 hour after patient transfer to postanesthesia care unit.
  The changes of glucagon and catecholamine during the surgery period
Effects of dexmedetomidine on perioperative cortisol (ng/ml) | before dexmedetomidine infusion, 1 hour after incision, at the end of surgery, 1 hour after patient transfer to postanesthesia care unit.
  The changes of cortisol during the surgery period

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China